CLINICAL TRIAL: NCT01166191
Title: Concurrent Chemo-radiotherapy With IMRT for Stage I-III Small Cell Lung Cancer
Brief Title: Concurrent Chemo-radiotherapy With Intensity-Modulated Radiation Therapy (IMRT) for Limited Disease Small Cell Lung Cancer (LD-SCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRONC 45.1,5
Record Dates: First submitted 2010-07-19; First posted 2010-07-20 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Stage I-III Small Cell Lung Cancer
Keywords: Radiotherapy; SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SCLC (Experimental)
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy

SUMMARY:
The investigators' group was the first to perform a phase II trial in patients with limited disease (stage I-III) small-cell lung carcinoma (SCLC) in which only the fluorodeoxyglucose-positron emission tomography (FDG-PET) positive lymph nodes were irradiated. In this trial, only 3% of isolated nodal failures were observed. However, all patients in that study were treated with 3D conformal radiotherapy (3DCRT). At present, IMRT techniques have become more standard in lung cancer. Because of the lower radiation dose to the lymph nodes outside of the planning target volume (PTV) with IMRT, higher incidences of isolated nodal failures may occur. In this trial, the investigators will investigate the patterns of local relapse after IMRT with concurrent chemotherapy in patients with stage I-III SCLC.

DETAILED DESCRIPTION:
Eligible patients (see below) will receive radiotherapy to the primary tumor and the initially involved mediastinal lymph nodes on FDG-PET scan to a dose of 45Gy in 30 fractions in 3 weeks (1.5Gy BID). Radiotherapy will be delivered concurrently with cisplatin (or in case of a creatinin clearance of <60ml/min, carboplatin) and etoposide chemotherapy. When after 4 cycles of chemotherapy and concurrent chest radiotherapy, no disease progression is observed and the WHO performance status is 0-2, PCI (prophylactic cranial irradiation) will bee offered to a dose of 25 Gy in 10 daily fractions.

The radiation doses will be specified according to ICRU 50. Lung density corrections will be applied, as well as all standard QA procedures. Technical requirements are the same as in standard practice at MAASTRO clinic.

ELIGIBILITY:
Inclusion Criteria:

* Histological of cytological proven SCLC
* UICC stage I-III, which are amendable for radical local treatment
* Performance status 0-2
* IMRT technique

Exclusion Criteria:

* Not SCLC or mixed SCLC and other histologies (e.g. non-small cell carcinoma)
* Stage IV
* Performance status 3 or more
* No IMRT technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Isolated nodal failures | 18 months
  Proportion of isolated nodal failures 18 months post-radiotherapy

SECONDARY OUTCOMES:
Progression-free survival | 18 months
Dyspnea (CTCAE 4.0) | 18 months
Dysphagia (CTCAE 4.0) | 18 months
Overall survival | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD, PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO clinic, Maastricht, Limburg, Netherlands